CLINICAL TRIAL: NCT04897412
Title: A 2-Stage Adaptive Design, Phase 2 Study to Evaluate the Efficacy, Safety and Tolerability of CBL-514 Injection for Reducing Abdominal and Thigh Subcutaneous Fat (Stage 2)
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of CBL-514 Injection for Reducing Subcutaneous Fat (Stage 2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Caliway Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBL-0202(Stage 2)
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Subcutaneous Fat

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBL-514 Injection (Experimental): Participant will receive CBL-514 administered in 2.4 mL injections, up to 120 mL per treatment session at intervals of approximately 4 weeks for up to a maximum of 4 treatments.
  Interventions: Drug: CBL-514 Injection
- Placebo: 0.9% Sodium Chloride (Placebo Comparator): Participant will receive 0.9% Sodium Chloride administered in 2.4 mL injections, up to 120 mL per treatment session at intervals of approximately 4 weeks for up to a maximum of 4 treatments.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CBL-514 Injection — Formulated as an injectable CBL-514 solution at a concentration of 5 mg/mL.
  Arms: CBL-514 Injection
Other: Placebo — Sodium Chloride (0.9% NaCl) placebo for injection
  Arms: Placebo: 0.9% Sodium Chloride

SUMMARY:
The Stage 2 of this phase 2 study will be a randomized, single-blind, placebo-controlled, parallel, and multiple-dose study to assess the efficacy, safety, and subject satisfaction of CBL-514.

DETAILED DESCRIPTION:
This is the 2nd stage of a 2-Stage adaptive design, phase 2 study to evaluate the efficacy, safety and tolerability of CBL- 514 injection for reducing abdominal subcutaneous fat. Stage 2 will be conducted as a single-blind, placebo-controlled study.

CBL-514 will be administered via injection into the subcutaneous adipose layer on abdomen. Each subject will receive up to 4 treatments of allocated CBL-514 (2 mg/cm2) or placebo administered on abdomen, once every 4 weeks and complete 2 follow-up visits after the last treatment. The maximum dose is 600 mg per treatment depending on the level of fat accumulation on subject's abdomen.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 years to 64 years old (at Screening), inclusive.
2. Body mass index (BMI) greater than 18.5 and less than 35 kg/m2 and body weight greater than or equal to 50 kg at Screening and Day 1.
3. Subject has subcutaneous fat thickness surrounding the center of localized area of treatment. For stage 2, abdominal skinfold thickness of at least 3.00 cm (30.0 mm) and up to 8.00 cm (80.0 mm) by pinch method (measured by calibrated caliper) at Screening.
4. Subject has stable body weight (identified as less than or equal to 5% weight change per subject report) for at least 3 months before Screening and during the study.
5. Subject who has maintained a stable lifestyle (e.g. exercise, eating patterns, and smoking habit) per subject report for at least 3 months before Screening and during the study.
6. Voluntarily signs the Informed Consent Form (ICF) and, in the opinion of the Investigator or delegate, is physically and mentally capable of participating in the study, and willing to adhere to study procedures.

Exclusion Criteria:

1. Female subject of childbearing potential who is not willing to commit to an acceptable contraceptive regimen with her partner from the time of Screening and throughout study participation until 90 days after the last IP dose, or who is currently pregnant or lactating. Male subject who is not willing to commit to an acceptable contraceptive method.

   Note: Subjects who are not of childbearing potential are not required to use contraception. Females with no childbearing potential are defined as who have been surgically sterilized (hysterectomy or bilateral oophorectomy) or who are post-menopausal (defined as at least 50 years with greater than or equal to 12 months of amenorrhea with a FSH greater than 40 IU/L).
2. Subject diagnosed with coagulation disorders or is receiving anticoagulant/antiplatelet therapy or medications or dietary supplements, which impede coagulation or platelet aggregation.
3. Subject has hemoglobin A1c (HbA1c) greater than or equal to 9%, delayed wound healing, or any diabetic risks which, in the opinion of Investigator, is inappropriate to participate in the study.
4. Subject has a clinically significant cardiovascular disease and abnormal findings in electrocardiogram (ECG).
5. Subject with active or prior history of malignancies within 5 years before Screening or being worked-up for a possible malignancy. Except adequately treated basal cell carcinoma of skin and in situ squamous cell carcinoma of skin would be eligible as per Investigator's discretion.
6. Subject with a history of human immunodeficiency virus (HIV)-1, infection or subjects with active HIV infection at Screening with positive HIV antigen/antibody (Ag/Ab) combo test.
7. Subject with a history of Trypanophobia, the extreme fear of medical procedures involving injections or needles, or who experience vasovagal syncope and faint or pass out at the sight of blood or a needle.
8. Subject has abnormal skin or local skin conditions at the treatment area, which in the opinion of Investigator, is inappropriate to participate in the study, including but not limited to any of the following:

   1. Skin manifestations of a systemic disease,
   2. Any abnormality of the skin or soft tissues of the area to be treated,
   3. Grade III cellulite (Nürnberger and Muller scale, Nürnberger F, 1978) at the area to be treated,
   4. Skin folding and fat folding on abdomen
   5. Sensory loss or dysesthesia in the area to be treated,
   6. Evidence of any cause of enlargement in the area to be treated other than localized abdominal or thigh subcutaneous fat,
   7. Tattoos on the area to be treated.
9. Subject who has undergone the following procedures:

   1. Previous surgery which caused scar tissues on the anticipated treatment area before Screening or during the study, except laparoscopic surgery and surgery which causes very small scar tissues would be eligible as per Investigator's discretion,
   2. Liposuction to the region to be treated before Screening or during the study,
   3. Esthetic procedure e.g. cryolipolysis, ultrasonic lipolysis, LLLT, lipolysis injection to the region to be treated within 12 months before Screening or during the study.
   4. Using medication which is delivered via subcutaneous injection at the treatment area during the study period.
10. Subject is on prescription or OTC weight reduction medication or weight reduction programs within 3 months before Screening or during the study.
11. Subject is undergoing chronic steroid or immunosuppressive therapy, with the exception of oral steroid inhalation indicated for asthma management or topical steroid application for skin conditions that are not directly applied or indirectly affect the treatment area.
12. Requiring continual use of the following therapeutic agents during the study: terfenadine (Teldane), buspirone (Buspar), fexofenadine (Fexotabs, Tefodine, Telfast, Xergic, Allegra, etc.), any medication that is known to strongly inhibit or induce CYP enzymes, sensitive CYP substrates or drugs with narrow therapeutic index, in the opinion of the investigator, may affect the evaluation of the study product or place the participant at undue risk.

    If a subject needs to use the above mentioned therapeutic agents during the study for any reason, these therapeutic agents should not be used at least for 2 days prior to dosing and until 1 day post-dose.
13. Unable to receive topical anesthesia (e.g., history of hypersensitivity to lidocaine).
14. Subjects with known allergies or sensitivities to the study treatment or its components.
15. Subjects with liver cirrhosis or with inadequate liver function at Screening defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALKP), total bilirubin (TBIL), or gamma-glutamyl transferase (GGT) greater than 3.0 × upper limit of normal (ULN), or with any hepatic medical condition that would interfere with assessment of safety or efficacy or compromise the subject's ability to undergo study procedures or provide informed consent.
16. Subjects with any renal impairment, defined as abnormal serum creatinine, and urea greater than 1.5 × ULN or estimated glomerular filtration rate (eGFR) less than 90 mL/min/1.73 m2. Subjects who are currently on dialysis should be excluded.

    Subjects with an eGFR greater than or equal to 60 and less than 90 mL/min/1.73 m2 at Screening should be evaluated by the Investigator to exclude pre-existing renal disease or associated dysfunction. If mild decrease in eGFR is assessed by the Investigator as not clinically significant or not related to dysfunction, the subjects may be eligible upon the Investigator's assessment.
17. Use of other investigational drug or device within 12 weeks prior to Screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who lose at least 150 mL of subcutaneous fat compared with placebo | From Visit 2 (Baseline) up to 8 weeks after last treatment
  The proportion of subjects who lose at least 150 mL of subcutaneous fat as measured by ultrasound from Baseline to follow-up visits compared with placebo.

SECONDARY OUTCOMES:
Proportion of subjects who lose at least 200 mL of subcutaneous fat compared with placebo | From Visit 2 (Baseline) up to 8 weeks after last treatment
  The proportion of subjects who lose at least 200 mL of subcutaneous fat as measured by ultrasound from Baseline to follow-up visits compared with placebo.
Number of treatments required to first occurrence of reducing at least 150 mL of subcutaneous fat volume in CBL-514 group | From Visit 2 (Baseline) up to 8 weeks after last treatment
  Evaluate the number of treatments required to first occurrence of reducing at least 150 mL of subcutaneous fat volume over the treated area as measured by ultrasound in CBL-514 group.
Change of subcutaneous fat volume over the treated area compared with placebo | From Visit 2 (Baseline) up to 8 weeks after last treatment
  Change of subcutaneous fat volume over the treated area as measured by ultrasound from Baseline to follow-up visits compared with placebo.
Change of subcutaneous fat volume over the treated area of the CBL-514 group compared with individual baseline | From Visit 2 (Baseline) up to 8 weeks after last treatment
  Change of subcutaneous fat volume over the treated area of the CBL-514 group as measured by ultrasound compared with individual Baseline.
Evaluation of safety following up to 4 courses of CBL-514 compared with placebo | Up to 8 weeks after last treatment
  Safety as assessed by recording of TEAEs, laboratory assessments, vital signs, ECGs, physical examinations, and ISRs compared with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sheu, Study Director — Caliway Biopharmaceuticals Co., Ltd.
Locations (5):
- United States (4):
  - Investigational site 1, Chicago, Illinois
  - Investigational site 2, Omaha, Nebraska
  - Investigational site 3, Nashville, Tennessee
  - Investigational site 4, Austin, Texas
- Investigational site 5, Melbourne, Victoria, Australia